CLINICAL TRIAL: NCT00252122
Title: A Pilot Study on the Effects of Intravenous Ketamine on Acute Pain Crisis in Patients With Sickle Cell Disease
Brief Title: Pilot Study on the Effects of Intravenous Ketamine on Acute Pain Crisis in Patients With Sickle Cell Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment was very slow.
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Arjunan Ganesh, MBBS, The Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-6-3708
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients receiving ketamine are those patients, arm 1, that are sill experiencing pain after Morphine has been given.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine. 0.2 mg/kg, intravenously
  Other Names: Ketalar

SUMMARY:
The purpose of this pilot study is to provide a preliminary assessment of the feasibility and efficacy of intravenous ketamine in controlling pain in patients with sickle cell disease (who are admitted to the hospital with severe, acute pain crisis, and who have been resistant to intravenous narcotics).

DETAILED DESCRIPTION:
It is often difficult to manage acute painful crisis in patients with sickle cell disease. The usual management of these crises relies on hydration, administration of oxygen and narcotics, like morphine. A select group of patients, for unknown reasons, does not respond to this management and these patients often require prolonged use (several days) of intravenous narcotics. Narcotics have proven to be ineffective in controlling this type of pain and can cause multiple side effects (sedation, vomiting, respiratory depression). We propose to administer intravenous ketamine in this group of patients who are resistant to intravenous narcotics. Ketamine has been proven to be effective in controlling pain in multiple clinical situations. However, there are no data in the literature describing its use in patients with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7 to <19
* Acute vaso-occlusive crisis
* Persistent pain despite initial pain management with intravenous (IV) opioids

Exclusion Criteria:

* Contraindications to the use of ketamine
* Mental retardation or psychological conditions that may affect the proper evaluation of pain and side effects
* Known allergy to ketamine

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2004-06; Primary Completion 2005-11 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Assessing pain scores within 48 hours after administration of the drug. Assessing decrease in pain and increase in mobility. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Arjunan Ganesh, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States